CLINICAL TRIAL: NCT07089576
Title: A Prospective, Multi-center Clinical Study to Evaluate the Safety and Effectiveness of Arcevo LSA in the Open Repair of Aortic Arch Aneurysms and Dissections
Brief Title: Clinical Study to Evaluate the Safety and Effectiveness of Arcevo LSA
Acronym: ARTIZEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artivion Inc. (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ART2401.000-C
Record Dates: First submitted 2025-07-17; First posted 2025-07-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Aortic Arch Aneurysm; Aortic Arch Dissection; Chronic Aortic Dissection; Acute Aortic Dissection
Keywords: total arch replacement; frozen elephant trunk; aortic arch aneurysm; aortic arch dissection
MeSH Terms: conditions — Aneurysm, Aortic Arch; Dissection, Thoracic Aorta

STUDY DESIGN:
Intervention Model Description: Primary Arm: chronic aortic dissection or aortic aneurysm. Secondary Arm: acute or subacute aortic dissection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Arcevo LSA (Experimental): The Primary study arm will consist of patients with an aortic aneurysm or chronic aortic dissection (n=117).
  The Secondary study arm will include patients with acute or subacute aortic dissections (n=15).
  Interventions: Device: Arcevo™ LSA Hybrid Stent Graft System

INTERVENTIONS:
Device: Arcevo™ LSA Hybrid Stent Graft System — The Arcevo LSA Hybrid Stent Graft System is an implantable aortic stent graft with LSA branch which is preloaded onto a delivery system and implanted during an open surgical procedure, or more specifically a total arch replacement procedure. The device is intended for use with a proximal surgical graft (not supplied). If additional coverage is needed, a protocol specified thoracic endovascular aortic repair (TEVAR) device may be used.

SUMMARY:
The goal of this clinical trial is to learn if the Arcevo LSA stent graft can safely and effectively treat patients that have an acute or chronic aortic dissection and/or aneurysm that involves the aortic arch and the descending thoracic aorta, with or without the involvement of the ascending aorta.

ELIGIBILITY:
General Inclusion Criteria

1. ≥18 years of age or ≤80 years of age (male or female) at time of surgery
2. Patient has one of the following indications for open surgery based on computed tomography angiography (CTA) completed within 90 days of informed consent:

   * Acute, subacute, or chronic dissection that involves the aortic arch and the descending thoracic aorta, with or without involvement of the ascending aorta
   * Aneurysm that involves the aortic arch and the descending thoracic aorta, with or without involvement of the ascending aorta
3. Patient, or patient's legally authorized representative (LAR; in the secondary arm only), provides written informed consent prior to any study procedures
4. Patient's surgery occurs within 90 days of informed consent

   Anatomical Inclusion Criteria
5. Aortic diameter at the intended Arcevo™ LSA anastomosis site is ≥ 21 mm
6. For Aneurysm with distal sealing (i.e., single stage procedure), aortic diameter at the intended distal sealing zone is between 20-36 mm
7. For Dissection with distal sealing, aortic diameter at the intended distal sealing zone is between 22-40 mm
8. LSA branch does not require additional stenting further into the LSA (beyond the Arcevo™ LSA)
9. The intended LSA sealing zone has a diameter between 8.5 mm and 14.0 mm with a length of at least 10 mm
10. Absence of dissection, aneurysm, or stenosis in the intended LSA sealing zone
11. The intended LSA branch position does not interrupt flow to any branch vessel (e.g., left vertebral artery)
12. Patient does not have computed tomography (CT) evidence of extreme arch or LSA angulation precluding safe passage of the Arcevo™ LSA and delivery system
13. LSA take-off angle between 15° and 90°
14. For patients requiring planned extension, there is a ≥ 2 cm distal seal zone for the TEVAR device without a severely angulated descending aorta
15. For patients requiring planned extension, patient has suitable iliac artery anatomy for safe passage of the TEVAR delivery system

General Exclusion Criteria

1. Patient is pregnant, or planning to become pregnant during the course of the study; individuals of child-bearing potential must agree to use acceptable methods of contraception during the study
2. Patient has another medical condition (aside from the arch disease) that, in the opinion of the investigator, reduces the patient's life expectancy to < 2 years
3. Patient has an existing aortic stent graft device in the descending aorta that would interact with Arcevo™ LSA
4. Patient has a medical, social, or psychological problem that, in the opinion of the investigator, could impede the patient's ability to return for follow-up
5. Patient is unwilling or unable to comply with the follow-up schedule
6. Patient is institutionalized due to administrative or judicial order
7. Patient is unwilling to accept blood transfusion or blood product
8. Patient is currently participating in another interventional clinical study which includes treatment with another investigational product (e.g., device, pharmaceutical or biologic)

   Medical Exclusion Criteria
9. Patient is unfit for open surgical repair involving circulatory arrest
10. Patient is in extreme hemodynamic compromise requiring cardiopulmonary resuscitation (CPR) or substantial inotropic support prior to surgery
11. Patient has an active systemic infection
12. Patient has endocarditis or active infection of the aorta
13. Patient has a freely ruptured aorta
14. Patient has a history of a bleeding disorder (e.g., hemophilia)
15. Patient has current end-stage renal disease (e.g., GFR <30 mL/min)
16. Patient has a known allergy to Arcevo™ LSA components and TEVAR device components (if required) (nitinol, polyester, platinum-iridium, or polyethylene)
17. Patient has uncontrollable anaphylaxis to iodinated contrast or other inability to obtain CT angiograms during follow-up
18. Patient has acute coronary malperfusion
19. Patient has symptomatic visceral malperfusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Composite Rate of Patients Free From ≥1 Major Adverse Event | 1 year post-index procedure of LSA stent graft implant
  The major adverse events included in the composite are:
  * All-cause mortality
  * New permanent disabling stroke
  * New permanent paraplegia and/or paraparesis
  * Unanticipated aortic reoperation in the treated segment
  * LSA occlusion

SECONDARY OUTCOMES:
Rate of Mortality | Follow-up at 30 days, 6, 12, 24, 36, 48, and 60 months of the index procedure
  All-cause, Cardiovascular-related, Aorta-related, Procedure-related, Device-related
Rate of Patients with ≥1 Additional Aortic Procedure | Follow-up at 30 days, 6, 12, 24, 36, 48, and 60 months of the index procedure
  All unplanned aortic procedures (endovascular, percutaneous, and open), Unanticipated aortic reoperations in the treated segment, Unanticipated device-related reoperations, Arcevo LSA explant
Rate of Patients with ≥1 Device-Related Event | Follow-up at 30 days, 6, 12, 24, 36, 48, and 60 months of the index procedure
  Device migration, Distal stent-induced new entry (d-SINE), Failed stent patency in the main body, Failed stent patency in the LSA, Stent-graft integrity issue compromising flow (i.e., stent fracture, narrowing, kink, or twist)
Rate of Patients with Major Adverse Events | Follow-up at 30 days, 6, 12, 24, 36, 48, and 60 months of the index procedure
  New permanent paraplegia, New permanent paraparesis, New temporary paraplegia, New disabling stroke, New non-disabling stroke, New transient ischemic attack, Aortic rupture, Bowel ischemia, Hypersensitivity, Myocardial infarction, New onset renal failure requiring temporary dialysis, New onset renal failure requiring permanent dialysis, Pseudoaneurysm, Recurrent laryngeal or phrenic nerve injury, Respiratory failure (need for reintubation or ventilator dependence >48 hours), Severe heart failure requiring mechanical circulatory support, Thromboembolic adverse events
Rate of Patients with Radiographic Events (determined by Core Lab) | Follow-up at 30 days, 6, 12, 24, 36, 48, and 60 months of the index procedure
  Anastomotic Leak between Arcevo™ LSA and surgical graft (i.e., Type Ia Endoleak or Distal anastomotic new entry [DANE]), Type Ic Endoleak (i.e. at the end of the LSA stent component), LSA occlusion, New LSA dissection, Maximal total aortic diameter growth >1 cm in the treated segment (Zones 2-4) compared to first post-operative CTA, Maximal total aortic diameter growth >1 cm at 1 cm beyond the distal end of Arcevo™ LSA, compared annually.
  Dissection Only:
  True lumen (TL) reduction compared to baseline > 5.0 mm at maximal total aortic diameter (Zones 2-4), False lumen (FL) growth compared to baseline > 5.0 mm at maximal total aortic diameter (Zones 2-4), FL thrombosis in the treated segment (LSA, Zones 2-4), FL thrombosis in the untreated segment (Zone 5).
Rate of Patients Requiring a Thoracic Extension Procedure who Experience Device-Extension Failure | Follow-up at 30 days, 6, 12, 24, 36, 48, and 60 months of the index procedure
  Any failure of device-extension integrity (e.g., wear or tear in the fabric or wire breakage) resulting in a compromised seal and blood leakage or movement of the device
Rate of Patient Requiring a Thoracic Extension Procedure with Evidence of Type IIIa Endoleak | Follow-up at 30 days, 6, 12, 24, 36, 48, and 60 months of index procedure
  Type IIIa Endoleak
Rate of Patients Requiring Thoracic Extension Procedure with Failed Patency | Follow-up at 30 days, 6, 12, 24, 36, 48, and 60 months of the index procedure
  Failed patency of the device-extension overlap
Rate of Patients Requiring Thoracic Extension Procedure with ≥1 Primary Major Adverse Events | 30 days post-extension procedure
  All-cause mortality, new permanent disabling stroke, new permanent paraplegia and/or paraparesis, unanticipated aortic reoperation in the treated segment, LSA occlusion
Rate of Patients Requiring Thoracic Extension Procedure Requiring ≥1 Secondary Procedure Related to Extension | 30 days post-extension procedure
  Secondary procedures related to the extension

OTHER OUTCOMES:
Rate of Patients with Technical Success | At exit from operating room
  Successful delivery and accurate placement of the device in the intended implantation site, as well as retrieval of the device delivery system, AND
  Patency of the device, including LSA, at conclusion of the procedure, AND
  No need for unanticipated or emergency surgery to correct a device malfunction or device-related complication
Rate of Patients with Procedural Success | At hospital discharge or at 30 days, whichever is longer at time of event
  Technical success with the absence of the following:
  Death,
  Major adverse ischemic events, including the following:
  New disabling stroke, New paraplegia, New paraparesis, New device-related ischemia (i.e., not evident at time of index procedure), Distal procedure-related thromboembolic adverse event.
  General procedure-related complications:
  New onset renal failure requiring dialysis, Bowel or limb ischemia requiring surgery or intervention, Additional unplanned surgical or interventional procedures related to the device, since completion of the index procedure
Rate of Patients with Treatment Success | Follow-up at 30 days, 6, 12, 24, 36, 48, and 60 months of the index procedure
  Technical success with the absence of the following:
  Aorta-related mortality.
  Major adverse ischemic events, including the following:
  New disabling stroke, New permanent paraplegia, New permanent paraparesis, Increase in total aortic diameter > 1.0 cm between scheduled post-operative imaging (performed per schedule of activities) in the treated region of the aorta (Zones 2-4), Aortic rupture, Fistula formation (i.e., aortobronchial or aortoenteric), Device-related occlusion of the aortic arch (Zones 2-4), Loss of device integrity (e.g., stent fracture that could affect fixation or seal, graft fabric hole or tear, collapse), New Type Ic endoleak.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Southern California, Los Angeles, California
  - Columbia University Irving Medical Center/New York Presbyterian Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Texas - Austin, Austin, Texas
  - Baylor Scott & White, Plano, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No